CLINICAL TRIAL: NCT06626425
Title: Smartphone-based Meditation Training to Reduce Adolescent Depression
Brief Title: Well-being Training for Adolescent Depressive Symptoms (TeenWell Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-0554; 1K01MH130752-01A1 (NIH); A483000 (Other: UW Madison); Protocol Version 5/22/25 (Other: UW Madison)
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-07

CONDITIONS: Depression
Keywords: adolescent; meditation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: This is a randomized active-controlled wait-list trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Healthy Minds Program (HMP) App (Experimental): The HMP is a smartphone meditation-based well-being training.
  Interventions: Other: Healthy Minds Program App
- Hydro Coach active control group (HC) (Active Comparator): The water tracking app is a publicly available, user-designed hydration app that prompts users to enter in daily liquid consumption and provides optimized hydration recommendations based on user input.
  Interventions: Other: Hydro Coach App

INTERVENTIONS:
Other: Healthy Minds Program App — An 8-week meditation-based well-being training containing content for each of the four pillars of the training program: Awareness, Connection, Insight, and Purpose.
  Arms: Healthy Minds Program (HMP) App
Other: Hydro Coach App — The Hydro Coach app (HC). A smartphone-based wellness app to ensure proper hydration.
  Arms: Hydro Coach active control group (HC)

SUMMARY:
This study is being done to see if the Healthy Minds Program app helps adolescents with elevated depressive symptoms. Up to 200 participants will be on study for 20 weeks.

DETAILED DESCRIPTION:
Participants will be randomized into one of two groups: Healthy Minds Program intervention group (HMP) or a water tracking active control group. The groups will use different mobile health apps for eight weeks. All participants will complete assessments pre-intervention, after weeks 2, 4, and 6 of the intervention, at week 8 (post-intervention), and at week 20 (follow-up). Participants will complete a short daily diary set of questions on their social interactions that day. Participants will wear a Biostrap band for continuous collection of heart rate, movement, and daily sleep indices, and geolocation data will be extracted from participant phones using the FollowMee app. Participants will receive access to the app they were not assigned to after follow-up.

Primary Objective

* Assess acceptability and preliminary efficacy of an 8-week mHealth meditation training program on depressive symptoms.

Secondary Objectives

* Investigate effects of the meditation training program on symptoms of anxiety, behavior (social isolation), psychophysiological processes related to health and disease (e.g., sleep). Test changes in behavior and psychophysiology as mechanisms of improved mental health. Test whether improved mental health is associated with improved academic outcomes.

ELIGIBILITY:
1. Age 14 to 19
2. Currently in high school (i.e., 9th to 12th grade) or if not attending school, would be in high school if enrolled
3. Proficient in English
4. Able to understand and provide informed consent (greater than or equal to 18 years old) or assent and parent/guardian consent (if less than 18 years old)
5. PROMIS Depression Scale T-score greater than or equal to 60
6. If on a psychotropic meditation, has been receiving a stable dose for greater than or equal to 4 weeks
7. Willing and able to complete all study procedures

Exclusion Criteria:

1. Has received a high school diploma or a high school equivalency diploma (HSED or GED)
2. Weekly or more frequent meditation practice
3. Prior use of the Healthy Minds Program app
4. Prior use of the water tracking app
5. Endorses current active suicidal ideation with intent on the baseline screen
6. Self-reported history of psychosis or mania
7. Practiced the techniques learned in a mindfulness-based therapy Acceptance Commitment Therapy (ACT), Dialectical Behavior Therapy (DBT), Mindfulness-Based Stress Reduction (MBSR) etc. one or more times per week in the last 6 months. Include therapy sessions if mindfulness is practiced in session or planning to start one of these therapies during the study period.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-07 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
PROMIS Pediatric Depression T-Scores | 8 weeks, 20 weeks
  Efficacy will be measured with the PROMIS Pediatric Item Bank (version 3.0) Depressive Symptoms Short Form 8a survey which results in T-scores where a score of less than 55 = None to slight depression, 55.0-59.9 = Mild depression, 60.0-69.9 = Moderate depression, 70 and over = Severe depression.

SECONDARY OUTCOMES:
PROMIS Pediatric Anxiety T-Scores | 8 weeks, 20 weeks
  T-score less than 55 = None to slight anxiety; between 55.0 and 59.9 = Mild anxiety; between 60.0 and 69.9 = Moderate anxiety; and 70 and over = Severe anxiety
EPOCH Wellbeing Scores | 8 weeks, 20 weeks
  The EPOCH Wellbeing score measures wellbeing in each of 4 domains: engagement, perseverance, optimism, and connectedness. It is scored on a 5 point likert scale from 1 (almost never) to 5 (almost always). Higher scores are indicative of increase wellbeing.
PROMIS Pediatric Sleep Disturbance T-Score | 8 weeks, 20 weeks
  T-score less than 55 = None to slight sleep disturbance; between 55.0 and 59.9 = Mild sleep disturbance; between 60.0 and 69.9 = Moderate sleep disturbance; and 70 and over = Severe sleep disturbance.
Sleep Duration assessed with wearable device | Daily through 20 weeks
  Total sleep time will be measured through the Biostrap device.
Sleep Staging assessed with wearable device | Daily through 20 weeks
  Proportion of sleep time awake, in REM and non-REM sleep will be measured through the Biostrap device and Philips sleep staging algorithm.
Wake after sleep onset | Daily through 20 weeks
  The amount of time awake after sleep onset will be assessed with the Biostrap device.
Pulse Rate Variability (PRV) collected by a wearable sensor | Daily through 20 weeks
  Root mean square of successive differences of heart beats and High-Frequency power will be analyzed.
Belonging Uncertainty Scale Score | 8 weeks, 20 weeks
  The Belonging Uncertainty Scale is scored from 1-7 where higher scores indicate more uncertainty about belonging.
Drexel Defusion Teen Score | 8 weeks, 20 weeks
  Drexel Defusion measures the ability to psychologically distance oneself internal thoughts and feelings. It is scored on a 6-point likert scale from 0 (not at all) to 5 (very much) for a total possible range of scores from 0-50, higher scores indicate increased ability to defuse.
NIH Toolbox - Emotional Battery Loneliness (Ages 8-17) Fixed Form | 8 weeks, 20 weeks
  The NIH Toolbox Loneliness pediatric scale is on a 5 point likert scale from 1 (never) to 5 (always) for a total range of scores from 7-35 where higher scores indicate increased feelings of loneliness.
Perseverative Thinking Questionnaire - Child Scores | 8 weeks, 20 weeks
  The Perseverative Thinking Questionnaire is scored on a 5 point likert scale, from 0 (never) to 4 (almost always) for a total possible range of scores from 0-60 where higher scores indicate increase repetitive negative thinking.
Healthy Minds Index | 8 weeks
  The Healthy Minds Index is a four factor measure of well-being that assesses skills in awareness, connection, insight and purpose. Each item is rated on a 1 (None of the time) to 5 (all of the time) scale, with higher scores representing greater endorsement of the construct. Subscale scores ranges from 4-30
Five Facet Mindfulness Questionnaire 16-item Adolescent version | 8 weeks
  A 16-item self-report that assesses four facets of mindfulness. Items are rated on a 0 (never or rarely true) to 5 (always true) scale, with higher scores representing greater mindfulness. Scores range from 0-80.
Attitudes Towards Online Psychological Interventions | 8 weeks
  A 4-item self-report rated on a 1 (strongly disagree) to 5 (strongly agree) scale that asks participants to report on their attitudes toward digital interventions. Higher scores reflect more positive attitudes. Scores range from 4-20.
Adverse Meditation Experience Questionnaire | 8 weeks, 20 weeks
  An 11-items self-report asking participants to note any difficulties they experience during meditation or attribute to meditation. Responses are coded quantitatively and qualitatively.

OTHER OUTCOMES:
Digital Working Alliance Inventory | Weeks 2, 4, 6, 8 and 20.
  A six-item inventory assessing the degree to which a participant feels alliance with a digital therapeutic. Scores ranges from 6 to 42, with higher scores representing greater alliance.
Growth mindset personality and intelligence | Baseline, week 8 and week 20.
  3-item scales assessing the degree to which a participant feels that their personality and intelligence are innate and unchanging or able to be affected by effort. Items are rated on 1 (Strongly disagree) to 6 (Strongly agree) scale, with higher scores (range 1-6) reflecting greater growth mindset.
Problematic Internet Use Scale | Baseline, week 8 and week 20
  A 3-item self-report inventory that asks participants to rate how often they feel negative effects of their technology use. Items are rated on a never(0) to very often (4) scale, with higher scores representing greater problematic internet use.
Daily diary of social interactions | Daily through 8 weeks
  A 1 to 6 item end of day experience sampling questionnaire assessing the presence, duration, quality and location of social interactions that day.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hirshberg, PhD, Principal Investigator — Center for Healthy Minds, UW Madison
Locations (1):
- Center for Healthy Minds, University of Wisconsin Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov, and results information from this trial will be submitted to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers 2 years after the completion of the primary endpoint by contacting the PI or accessing the data on osf.io.